CLINICAL TRIAL: NCT02481830
Title: An Open-label, Randomized, Phase 3 Study of Nivolumab or Chemotherapy in Subjects With Relapsed Small-cell Lung Cancer After Platinum-based First Line Chemotherapy (CheckMate 331: CHECKpoint Pathway and nivoluMAb Clinical Trial Evaluation 331)
Brief Title: Effectiveness Study of Nivolumab Compared to Chemotherapy in Patients With Relapsed Small-cell Lung Cancer
Acronym: CheckMate331
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Collaborators: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA209-331; 2015-001097-18 (EudraCT Number)
Record Dates: First submitted 2015-06-23; First posted 2015-06-25 (Estimated); Results first posted 2020-01-09 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Nivolumab; Topotecan; amrubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A Nivolumab (Experimental): Nivolumab intravenous infusion as specified
  Interventions: Drug: Nivolumab
- Arm B Chemotherapy Topotecan (Active Comparator): Topotecan as specified
  Interventions: Drug: Topotecan
- Arm B Chemotherapy Amrubicin (Active Comparator): Amrubicin intravenous infusion as specified (upon investigator's choice, where locally approved for 2nd line SCLC treatment)
  Interventions: Drug: Amrubicin

INTERVENTIONS:
Drug: Nivolumab
  Arms: Arm A Nivolumab
Drug: Topotecan
  Arms: Arm B Chemotherapy Topotecan
Drug: Amrubicin
  Arms: Arm B Chemotherapy Amrubicin

SUMMARY:
The purpose of this study is to compare the overall survival of nivolumab versus chemotherapy in subjects with relapsed SCLC.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed small cell lung cancer (SCLC)
* Subjects with either limited or extensive disease stage at the initial diagnosis
* Must have recurrence or progression after platinum-based first-line chemotherapy or chemoradiation therapy for the treatment of limited or extensive disease stage SCLC
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1

Exclusion Criteria:

* Untreated or symptomatic central nervous system (CNS) metastases
* Prior therapy with anti-PD-1, anti-PDL1, anti-PD-L2, anti-CD137, or anti-CTLA-4 antibody
* Inadequate hematologic or hepatic function

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 569 (Actual)
Dates: Start 2015-09-14 (Actual); Primary Completion 2018-08-17 (Actual); Study Completion 2022-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (151):
- United States (14):
  - Local Institution - 0065, Little Rock, Arkansas
  - Local Institution - 0024, New Haven, Connecticut
  - Local Institution - 0018, Atlanta, Georgia
  - Local Institution - 0056, St Louis, Missouri
  - Local Institution - 0088, Lincoln, Nebraska
  - Local Institution - 0173, Johnson City, New York
  - Local Institution - 0001, Durham, North Carolina
  - Local Institution - 0090, Cleveland, Ohio
  - Local Institution - 0002, Bethlehem, Pennsylvania
  - Local Institution - 0057, Lancaster, Pennsylvania
  - Local Institution - 0053, Philadelphia, Pennsylvania
  - Local Institution - 0089, Nashville, Tennessee
  - Local Institution - 0009, Nashville, Tennessee
  - Local Institution - 0070, Kennewick, Washington
- Australia (6):
  - Local Institution - 0102, Waratah, New South Wales
  - Local Institution - 0030, Brisbane, Queensland
  - Local Institution - 0031, Elizabeth Vale, South Australia
  - Local Institution - 0103, Kurralta Park, South Australia
  - Local Institution - 0028, Perth, Western Australia
  - Local Institution - 0027, Murdoch
- Austria (3):
  - Local Institution - 0085, Graz
  - Local Institution - 0086, Vienna
  - Local Institution - 0084, Wels
- Belgium (4):
  - Local Institution - 0013, Brussels
  - Local Institution - 0012, Edegem
  - Local Institution - 0011, Leuven
  - Local Institution - 0010, Yvoir
- Brazil (4):
  - Local Institution - 0095, Ijuí, Rio Grande do Sul
  - Local Institution - 0094, Porto Alegre, Rio Grande do Sul
  - Local Institution - 0093, Barretos, São Paulo
  - Local Institution - 0099, São Paulo
- Local Institution - 0025, Recoleta, Santiago de Chile, Chile
- China (17):
  - Local Institution - 0200, Beijing, Beijing Municipality
  - Local Institution - 0199, Beijing, Beijing Municipality
  - Local Institution - 0188, Beijing, Beijing Municipality
  - Local Institution - 0190, Beijing, Beijing Municipality
  - Local Institution - 0197, Guanzhou, Guangdong
  - Local Institution - 0189, Zhengzhou, Henan
  - Local Institution - 0194, Nanjing, Jiangsu
  - Local Institution - 0187, Changchun, Jilin
  - Local Institution - 0186, Xi'an, Shaanxi
  - Local Institution - 0181, Shanghai, Shanghai Municipality
  - Local Institution - 0185, Shanghai, Shanghai Municipality
  - Local Institution - 0202, Ürümqi, Xinjiang
  - Local Institution - 0183, Hangzhou, Zhejiang
  - Local Institution - 0201, Beijing
  - Local Institution - 0198, Guangzhou
  - Local Institution - 0182, Hangzhou
  - Local Institution - 0192, Shanghai
- Czechia (4):
  - Local Institution - 0069, Brno
  - Local Institution - 0067, Brno
  - Local Institution - 0068, Olomouc
  - Local Institution - 0066, Prague
- Denmark (3):
  - Local Institution - 0106, Copenhagen
  - Local Institution - 0098, Herlev
  - Local Institution - 0100, Odense
- France (6):
  - Local Institution - 0134, Brest
  - Local Institution - 0116, Lille
  - Local Institution - 0118, Paris
  - Local Institution - 0131, Pringy
  - Local Institution - 0132, Reims
  - Local Institution - 0117, Toulon
- Germany (15):
  - Local Institution - 0061, Bamberg
  - Local Institution - 0055, Berlin
  - Local Institution - 0023, Cologne
  - Local Institution - 0047, Essen
  - Local Institution - 0071, Frankfurt am Main
  - Local Institution - 0060, Gera
  - Local Institution - 0019, Gerlingen
  - Local Institution - 0021, Großhansdorf
  - Local Institution - 0058, Halle
  - Local Institution - 0059, Hamburg
  - Local Institution - 0020, Heidelberg
  - Local Institution - 0046, Immenstadt im Allgäu
  - Local Institution - 0022, München
  - Local Institution - 0054, Oberhausen
  - Local Institution - 0064, Regensburg
- Greece (3):
  - Local Institution - 0063, Heraklion, Crete
  - Local Institution - 0062, Athens
  - Local Institution - 0097, Thessaloniki
- Hungary (3):
  - Local Institution - 0112, Budapest
  - Local Institution - 0110, Budapest
  - Local Institution - 0150, Budapest
- Israel (4):
  - Local Institution - 0139, Beersheba
  - Local Institution - 0138, Kfar Saba
  - Local Institution - 0136, Ramat Gan
  - Local Institution - 0166, Safed
- Italy (8):
  - Local Institution - 0081, Bologna
  - Local Institution - 0073, Livorno
  - Local Institution - 0108, Lucca
  - Local Institution - 0077, Meldola
  - Local Institution - 0078, Milan
  - Local Institution - 0080, Monza
  - Local Institution - 0107, Rimini
  - Local Institution - 0079, Roma
- Japan (20):
  - Local Institution - 0169, Nagoya, Aichi-ken
  - Local Institution - 0159, Nagoya, Aichi-ken
  - Local Institution - 0196, Kashiwa, Chiba
  - Local Institution - 0155, Matsuyama, Ehime
  - Local Institution - 0153, Fukuoka, Fukuoka
  - Local Institution - 0168, Akashi-shi, Hyōgo
  - Local Institution - 0163, Kobe, Hyōgo
  - Local Institution - 0164, Natori-shi, Miyagi
  - Local Institution - 0161, Niigata, Niigata
  - Local Institution - 0171, Habikino-shi, Osaka
  - Local Institution - 0175, Hirakata-shi, Osaka
  - Local Institution - 0165, Osaka, Osaka
  - Local Institution - 0151, Ōsaka-sayama, Osaka
  - Local Institution - 0160, Sakai, Osaka
  - Local Institution - 0162, Kitaadachi-gun, Saitama
  - Local Institution - 0176, Bunkyo-ku, Tokyo
  - Local Institution - 0170, Chuo-ku, Tokyo
  - Local Institution - 0174, Chuo-ku, Tokyo
  - Local Institution - 0152, Wakayama, Wakayama
  - Local Institution - 0154, Tokyo
- Norway (2):
  - Local Institution - 0096, Bergen
  - Local Institution - 0072, Oslo
- Poland (6):
  - Local Institution - 0044, Elblag
  - Local Institution - 0041, Gdansk
  - Local Institution - 0032, Krakow
  - Local Institution - 0033, Lodz
  - Local Institution - 0042, Poznan
  - Local Institution - 0035, Warsaw
- Romania (4):
  - Local Institution - 0135, Bucharest
  - Local Institution - 0114, Craiova
  - Local Institution - 0113, Romania
  - Local Institution - 0149, Timisoara, Timis
- Russia (4):
  - Local Institution - 0122, Moscow
  - Local Institution - 0121, Ryazan
  - Local Institution - 0119, Saint Petersburg
  - Local Institution - 0126, Saint Petersburg
- South Korea (4):
  - Local Institution - 0145, Suwon, Gyeonggi-do
  - Local Institution - 0146, Cheongju-si
  - Local Institution - 0147, Seoul
  - Local Institution - 0148, Seoul
- Spain (6):
  - Local Institution - 0006, Barcelona
  - Local Institution - 0005, Barcelona
  - Local Institution - 0004, Madrid
  - Local Institution - 0003, Madrid
  - Local Institution - 0008, Seville
  - Local Institution - 0007, Valencia
- Switzerland (4):
  - Local Institution - 0104, Basel
  - Local Institution - 0133, Lausanne
  - Local Institution - 0109, Winterthur
  - Local Institution - 0156, Zurich
- Local Institution - 0143, Taichung, Taiwan
- United Kingdom (5):
  - Local Institution - 0157, London, Greater London
  - Local Institution - 0082, Manchester, Greater Manchester
  - Local Institution - 0083, Maidstone, Kent
  - Local Institution - 0124, Sutton, Surrey
  - Local Institution - 0123, Southampton

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — http://www.BMSStudyConnect.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Group A: Nivolumab 240mg IV on Day 1 of a 14-day cycle
- Group B: Chemotherapy (Topotecan 1.5 mg/m^2 IV or 2.3 mg/m^2 oral once daily on Days 1 to 5 of a 21-day cycle / Amrubicin 40 mg/m^2 IV once daily on Days 1 to 3 of a 21-day cycle)
Period: Pre-treatment
Arm/Group | Group A | Group B
Started (Randomized) | 284 | 285
Completed (Treated) | 282 | 265
Not Completed | 2 | 20
Not completed — Participant no longer meets Study Criteria | 1 | 4
Not completed — Withdrawal by Subject | 0 | 10
Not completed — Disease Progression | 1 | 1
Not completed — Other reasons | 0 | 1
Not completed — Participant request to discontinue study treatment | 0 | 4
Period: Treatment
Arm/Group | Group A | Group B
Started (Treated) | 282 | 265
Completed | 0 | 0
Not Completed | 282 | 265
Not completed — Disease Progression | 233 | 171
Not completed — Study drug toxicity | 18 | 38
Not completed — Death | 1 | 1
Not completed — Adverse Event unrelated to Study drug | 14 | 11
Not completed — Participants request to discontinue Study treatment | 6 | 34
Not completed — Withdrawal by Subject | 2 | 3
Not completed — Lost to Follow-up | 1 | 0
Not completed — Maximum Clinical Benefit | 0 | 5
Not completed — Administrative reason by sponsor | 1 | 1
Not completed — Other reasons | 6 | 1

BASELINE CHARACTERISTICS:
Population: All Randomized Participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Total
Number analyzed (Participants) | 284 | 285 | 569
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.5 (9.2) | 61.6 (8.4) | 61.6 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 110 | 108 | 218
  Male | 174 | 177 | 351
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 6 | 10
  Not Hispanic or Latino | 125 | 142 | 267
  Unknown or Not Reported | 155 | 137 | 292
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 70 | 71 | 141
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 211 | 211 | 422
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: The time from randomization to the date of death, data was based on Kaplan-Meier Estimates. A participant who has not died will be censored at last known date alive.
Time Frame: OS was followed continuously while participants were on the study drug and every 3 months, minimum follow up for overall survival was 15.8 months
Population: All Randomized Participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Group A | Group B
Number analyzed (Participants) | 284 | 285
Months | 7.46 [5.65 to 9.20] | 8.38 [7.03 to 10.02]
Statistical Analysis 1: Comparison: Group A vs Group B; Test type: Superiority; p = 0.1144, Log Rank; Hazard Ratio (HR) = 0.86, 95% CI 2-sided [0.72 to 1.04] — Stratified Cox proportional hazard model. Hazard Ratio is Nivolumab over Topotecan/Amrubicin

2. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS is defined as the time from randomization to the date of the first documented tumor progression based on investigator assessment (per RECIST 1.1), or death due to any cause. Participants who die without a reported prior progression will be considered to have progressed on the date of their death. Participants who did not progress or die will be censored on the date of their last evaluable tumor assessment. Participants who did not have any on study tumor assessments and did not die will be censored on the date they were randomized. Participants who started any subsequent anti-cancer therapy without a prior reported progression will be censored at the last evaluable tumor assessment prior to initiation of the subsequent anti-cancer therapy.
  Progressive disease (PD)= At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. The sum must demonstrate an absolute increase of at least 5 mm.
Time Frame: From randomization to the date of first documented tumor progression, or death due to any cause. Tumor response assessed every 6 weeks from first dose until week 30, and every 12 weeks (Up to approximately 80 months)
Population: All Randomized Participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Group A | Group B
Number analyzed (Participants) | 284 | 285
Months | 1.45 [1.41 to 1.51] | 3.71 [2.96 to 4.24]
Statistical Analysis 1: Comparison: Group A vs Group B; Test type: Superiority; Hazard Ratio (HR) = 1.39, 95% CI 2-sided [1.16 to 1.66] — Hazard Ratio is Nivolumab over Topotecan/Amrubicin using Stratified Cox proportional hazard model

3. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR is defined as the percentage of randomized participants whose best overall response (BOR) from baseline is either a complete response (CR) or partial response (PR) based on investigator assessment per RECIST 1.1 criteria. For participants without documented progression or subsequent anti-cancer therapy, all available response designations will contribute to the BOR determination. For participants who continue nivolumab beyond progression, the BOR should be determined based on tumor assessments before initial RECIST 1.1 defined progression.
  CR= Disappearance of all target lesions. Any pathological lymph nodes must have reduction in short axis to <10 mm.
  PR= At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
  Progressive disease (PD)= At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. The sum must demonstrate an absolute increase of at least 5 mm.
Time Frame: From randomization to the date of objectively documented progression or the date of subsequent anti-cancer therapy, whichever occurs first (Up to approximately 80 months)
Population: All Randomized Participants
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Group A | Group B
Number analyzed (Participants) | 284 | 285
Percentage of Participants | 13.7 [10.0 to 18.3] | 16.8 [12.7 to 21.7]
Statistical Analysis 1: Comparison: Group A vs Group B; Test type: Superiority; Estimate of Odds Ratio (OR) = 0.78, 95% CI 2-sided [0.49 to 1.24] — Strata adjusted odds ratio (Nivolumab over Topotecan/Amrubicin) using Mantel-Haenszel method

4. Post Hoc Outcome: Overall Survival (OS) - Extended Collection
Description: as for outcome 1
Time Frame: OS was followed continuously while participants were on the study drug and every 3 months, minimum follow up for overall survival was 64 months (Up to approximately 80 months)
Population: All Randomized Participants
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Group A | Group B
Number analyzed (Participants) | 284 | 285
Months | 7.46 [5.65 to 9.20] | 8.38 [7.03 to 10.02]
Statistical Analysis 1: Comparison: Group A vs Group B; Test type: Superiority; Hazard Ratio (HR) = 0.87, 95% CI 2-sided [0.73 to 1.04] — Stratified Cox proportional hazard model. Hazard Ratio is Nivolumab over Topotecan/Amrubicin

ADVERSE EVENTS:
Time Frame: SAEs and Other AEs are assessed from first dose to 100 days post last dose (Up to approximately 72 months). Participants were assessed for all-cause mortality from their randomization to study completion (Up to approximately 80 months).
Description: The number at Risk for All-Cause Mortality represents all Randomized Participants. The number at Risk for Serious Adverse Events and Other (Not Including Serious) Adverse Events represents all participants that received at least 1 dose of study medication.
Arm/Group | Group A | Group B
All-Cause Mortality (participants affected / at risk) | 251/284 | 256/285
Serious Adverse Events (participants affected / at risk) | 183/282 | 171/265
Other Adverse Events (participants affected / at risk) | 249/282 | 248/265
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group A (N=282) | Group B (N=265)
Anaemia (Blood and lymphatic system disorders) | 3 | 14
Bone marrow failure (Blood and lymphatic system disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 7 | 23
Leukopenia (Blood and lymphatic system disorders) | 1 | 3
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1
Myelosuppression (Blood and lymphatic system disorders) | 0 | 10
Neutropenia (Blood and lymphatic system disorders) | 0 | 11
Pancytopenia (Blood and lymphatic system disorders) | 0 | 8
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 15
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 1
Atrial flutter (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 2 | 1
Cardiac failure acute (Cardiac disorders) | 1 | 0
Cardiac tamponade (Cardiac disorders) | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1
Adrenocorticotropic hormone deficiency (Endocrine disorders) | 1 | 0
Cushing's syndrome (Endocrine disorders) | 1 | 0
Hyperthyroidism (Endocrine disorders) | 2 | 0
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1 | 2
Secondary adrenocortical insufficiency (Endocrine disorders) | 0 | 1
Abdominal hernia obstructive (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 4 | 4
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 2 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 4 | 1
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Immune-mediated enterocolitis (Gastrointestinal disorders) | 1 | 0
Intestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 2
Oral disorder (Gastrointestinal disorders) | 1 | 0
Small intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 1
Asthenia (General disorders) | 0 | 5
Chest pain (General disorders) | 1 | 0
Death (General disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
General physical health deterioration (General disorders) | 8 | 6
Malaise (General disorders) | 1 | 1
Mucosal inflammation (General disorders) | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 1
Oedema peripheral (General disorders) | 1 | 0
Pain (General disorders) | 1 | 2
Performance status decreased (General disorders) | 0 | 1
Pyrexia (General disorders) | 4 | 3
Sudden death (General disorders) | 0 | 1
Drug-induced liver injury (Hepatobiliary disorders) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 0
Hepatitis (Hepatobiliary disorders) | 1 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0
Bacteraemia (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 2 | 0
Bronchitis bacterial (Infections and infestations) | 1 | 0
Bullous erysipelas (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1
Chronic sinusitis (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 0 | 1
Encephalitis (Infections and infestations) | 1 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 1
Erysipelas (Infections and infestations) | 0 | 1
Herpes simplex (Infections and infestations) | 1 | 0
Infectious pleural effusion (Infections and infestations) | 1 | 0
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1 | 0
Localised infection (Infections and infestations) | 0 | 1
Neutropenic sepsis (Infections and infestations) | 0 | 4
Ophthalmic herpes zoster (Infections and infestations) | 0 | 1
Peritonsillar abscess (Infections and infestations) | 1 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 15 | 9
Pneumonia aspiration (Infections and infestations) | 1 | 0
Pneumonia bacterial (Infections and infestations) | 1 | 0
Post procedural infection (Infections and infestations) | 0 | 1
Pulmonary sepsis (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 3 | 2
Sepsis (Infections and infestations) | 2 | 2
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 2 | 1
Vascular device infection (Infections and infestations) | 0 | 2
Bone contusion (Injury, poisoning and procedural complications) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 1
Injection related reaction (Injury, poisoning and procedural complications) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Synovial rupture (Injury, poisoning and procedural complications) | 0 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | 0
Amylase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 1 | 0
Blood electrolytes abnormal (Investigations) | 0 | 1
C-reactive protein increased (Investigations) | 0 | 2
Gamma-glutamyltransferase increased (Investigations) | 1 | 0
Lipase increased (Investigations) | 2 | 0
Neutrophil count decreased (Investigations) | 2 | 4
Platelet count decreased (Investigations) | 4 | 10
White blood cell count decreased (Investigations) | 1 | 2
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 1
Glucose tolerance impaired (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 5 | 3
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoporotic fracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 1
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Epiglottic cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 108 | 85
Pericardial effusion malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Second primary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma of the tongue (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tongue neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour invasion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Brain oedema (Nervous system disorders) | 1 | 0
Cerebellar ataxia (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 2
Epilepsy (Nervous system disorders) | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 1
Hemiparesis (Nervous system disorders) | 0 | 1
Lacunar infarction (Nervous system disorders) | 1 | 0
Neurological symptom (Nervous system disorders) | 0 | 1
Paraneoplastic neurological syndrome (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 1 | 0
Spinal cord compression (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Toxic encephalopathy (Nervous system disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 2 | 2
Delirium (Psychiatric disorders) | 0 | 1
Disorientation (Psychiatric disorders) | 0 | 1
Bladder dilatation (Renal and urinary disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 2
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 | 8
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Mediastinal disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oesophagobronchial fistula (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 10 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0
Paraneoplastic pemphigus (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0
Poor venous access (Vascular disorders) | 0 | 1
Shock (Vascular disorders) | 0 | 1
Superior vena cava syndrome (Vascular disorders) | 0 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Group A (N=282) | Group B (N=265)
Anaemia (Blood and lymphatic system disorders) | 68 | 163
Leukopenia (Blood and lymphatic system disorders) | 12 | 41
Neutropenia (Blood and lymphatic system disorders) | 17 | 93
Thrombocytopenia (Blood and lymphatic system disorders) | 19 | 78
Hypothyroidism (Endocrine disorders) | 23 | 1
Abdominal pain (Gastrointestinal disorders) | 19 | 14
Abdominal pain upper (Gastrointestinal disorders) | 16 | 11
Constipation (Gastrointestinal disorders) | 45 | 49
Diarrhoea (Gastrointestinal disorders) | 34 | 44
Nausea (Gastrointestinal disorders) | 48 | 59
Stomatitis (Gastrointestinal disorders) | 12 | 17
Vomiting (Gastrointestinal disorders) | 33 | 41
Asthenia (General disorders) | 65 | 60
Fatigue (General disorders) | 63 | 78
Oedema peripheral (General disorders) | 12 | 17
Pyrexia (General disorders) | 28 | 37
Pneumonia (Infections and infestations) | 16 | 22
Upper respiratory tract infection (Infections and infestations) | 15 | 13
Infusion related reaction (Injury, poisoning and procedural complications) | 8 | 16
Alanine aminotransferase increased (Investigations) | 22 | 13
Amylase increased (Investigations) | 15 | 2
Aspartate aminotransferase increased (Investigations) | 22 | 16
Blood alkaline phosphatase increased (Investigations) | 16 | 9
Gamma-glutamyltransferase increased (Investigations) | 20 | 11
Haemoglobin decreased (Investigations) | 5 | 14
Lipase increased (Investigations) | 27 | 4
Neutrophil count decreased (Investigations) | 28 | 60
Platelet count decreased (Investigations) | 20 | 63
Weight decreased (Investigations) | 26 | 16
White blood cell count decreased (Investigations) | 26 | 46
Decreased appetite (Metabolism and nutrition disorders) | 79 | 70
Hyperglycaemia (Metabolism and nutrition disorders) | 15 | 8
Hypokalaemia (Metabolism and nutrition disorders) | 19 | 18
Hyponatraemia (Metabolism and nutrition disorders) | 24 | 25
Arthralgia (Musculoskeletal and connective tissue disorders) | 27 | 17
Back pain (Musculoskeletal and connective tissue disorders) | 30 | 25
Pain in extremity (Musculoskeletal and connective tissue disorders) | 16 | 11
Dizziness (Nervous system disorders) | 20 | 17
Headache (Nervous system disorders) | 30 | 21
Insomnia (Psychiatric disorders) | 23 | 17
Cough (Respiratory, thoracic and mediastinal disorders) | 63 | 52
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 63 | 45
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 15
Productive cough (Respiratory, thoracic and mediastinal disorders) | 20 | 8
Alopecia (Skin and subcutaneous tissue disorders) | 4 | 26
Pruritus (Skin and subcutaneous tissue disorders) | 27 | 4
Rash (Skin and subcutaneous tissue disorders) | 21 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (2):
  • Study Protocol (2018-03-20): https://cdn.clinicaltrials.gov/large-docs/30/NCT02481830/Prot_002.pdf
  • Statistical Analysis Plan (2018-08-14): https://cdn.clinicaltrials.gov/large-docs/30/NCT02481830/SAP_001.pdf